CLINICAL TRIAL: NCT03343119
Title: Transfer Routes of Antibiotic Resistance
Brief Title: Epidemiology of Resistant Microbial Strains Among Different Groups of People (Healthy, Infected and Exposed to Animals)
Acronym: ABRESIST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University of Tartu (Other)
Collaborators: Estonian University of Life Sciences (Other)
Responsible Party: Principal Investigator, Kaidi Telling, MD, University of Tartu
Other Study IDs: SLOTI12038T
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: ESBL Producing E.Coli; ESBL Producing K.Pneumoniae; Multidrug Resistant P.Aeruginosa; Carbapenem Resistant P.Aeruginosa; Methicillin Resistant Staphylococcus Aureus (MRSA); Vancomycin (Glycopeptide) Resistant Enterococcus (VRE)

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Other
Biospecimen Retention: Samples With DNA — DNA from isolated multiresistant bacteria
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Hospitalised patients: No intervention
- Healthy volunteers: No intervention
- Dog owners (healthy volunteers): No intervention
- Veterinarians (healthy volunteers): No intervention
- Pig farmers (healthy volunteers): No intervention

SUMMARY:
This study investigates carriage rate and risk factors for acquiring multiresistant bacteria (ESBL producing E.coli and K.pneumoniae, carbapenem-resistant and multidrug resistant P.aeruginosa, MRSA and VRE) in hospitalised patients and healthy volunteers.

ELIGIBILITY:
I group Hospitalised patients Inclusion Criteria

* MDR bacteria (listed above) isolated from clinical specimen
* hospitalisation to the Tartu University Hospital or North Estonia Medical Centre or West Tallinn Central Hospital or East-Tallinn Central Hospital or The Hospital of Reconstructive Surgery

II group Healthy volunteers Inclusion Criteria

* age >6 months
* have not received any antibacterial treatment in previous 3 months
* have not been hospitalised in previous 3 months

III group Dog owners Inclusion Criteria

* age >6 months
* have not received any antibacterial treatment in previous 3 months
* have not been hospitalised in previous 3 months
* owning a dog

IV group veterinarians Inclusion Criteria

* have not received any antibacterial treatment in previous 3 months
* have not been hospitaliZed in previous 3 months
* working as a veterinarian

V group pig farmers Inclusion Criteria

* have not received any antibacterial treatment in previous 3 months
* have not been hospitalized in previous 3 months
* occupation as a pig farmer

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: I group All individuals who have been hospitalised and have been diagnosed carriage or infection with multiresistant bacteria listed above.
  II group Children >6 months of age and all adults who have not been hospitalised or received antibacterial treatment in previous 3 months.
Sampling Method: Probability Sample
Enrollment: 708 (Actual)
Dates: Start 2012-03-27 (Actual); Primary Completion 2014-01-30 (Actual); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Colonization rate with multiresistant (MDR) bacteria in hospitalized patients | March 2012 - March 2014
  To evaluate the impact of hospitalization for carriage and infection rate with MDR bacteria
Colonization rate with multiresistant (MDR) bacteria in healthy humans | March 2012 - March 2014
  To evaluate the impact of animal exposure for carriage rate with MDR bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Tanel Tenson, PhD, Study Director — University of Tartu

REFERENCES:
- [Derived] Telling K, Laht M, Brauer A, Remm M, Kisand V, Maimets M, Tenson T, Lutsar I. Multidrug resistant Pseudomonas aeruginosa in Estonian hospitals. BMC Infect Dis. 2018 Oct 11;18(1):513. doi: 10.1186/s12879-018-3421-1. PMID 30309321